CLINICAL TRIAL: NCT04178031
Title: Association Between Clinical,Laboratory,Ultrasongraphy Predictors And Development of Copper IUD Complications
Brief Title: Association Between Clinical, Laboratory, Ultrasongraphy Predictors And Development of Copper IUD Complications
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed M Maged, MD, professor, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 172
Record Dates: First submitted 2019-11-24; First posted 2019-11-26 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: Intrauterine Device Migration
MeSH Terms: conditions — Intrauterine Device Migration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IUD insertion group (Experimental): All participants will have IUD inserted and follow up for occurance of complications
  Interventions: Device: IUD insertion

INTERVENTIONS:
Device: IUD insertion — Insert a warm, moistened speculum. Cleanse the cervix with an antiseptic solution. Apply gentle traction with the tenaculum to straighten the canal. Remove the sound by its handle and gently insert to measure the depth of the uterus. Do not apply great force if there is resistance. Apply further traction to the tenaculum and attempt to re-insert the sound at a different angle. Once the sound is inserted and removed, note the depth of the uterine cavity. The woman can expect to feel cramping as the sound is inserted and withdrawn.
  Load the IUD and insert it into the uterine cavity according to the manufacturer instructions. As the IUD is inserted through the cervix into the uterus, the patient may have pain and cramping similar to strong menstrual cramps.
  Gently remove the tenaculum. Trim the strings of the IUD to 3-4 cm in length Remove the speculum and assess the woman.

SUMMARY:
Only clinicians with proven proficiency in IUD insertion will be allowed to perform insertions . The steps of the IUD insertion procedure will be explained to the woman.

Perform a bimanual examination to determine the size, shape, and position of the uterus.

Insert a warm, moistened speculum. Cleanse the cervix with an antiseptic solution using 3 scoppettes or more (one for each sweep of the cervix).

Open the sterile insertion instruments without touching the inside of the packet and place within easy reach.

Remove the tenaculum by its handle and grasp the anterior or posterior lip of the cervix. Close gently to the first notch. Having the woman to cough while the tenaculum is being attached can ease the pinch.

Apply gentle traction with the tenaculum to straighten the canal. Remove the sound by its handle and gently insert to measure the depth of the uterus. Do not apply great force if there is resistance. Apply further traction to the tenaculum and attempt to re-insert the sound at a different angle. Once the sound is inserted and removed, note the depth of the uterine cavity. The woman can expect to feel cramping as the sound is inserted and withdrawn.

Open the IUD pack without touching its contents. Put on sterile gloves. Load the IUD and insert it into the uterine cavity according to the manufacturer instructions. As the IUD is inserted through the cervix into the uterus, the patient may have pain and cramping similar to strong menstrual cramps.

Gently remove the tenaculum. Tamponade any bleeding from the tenaculum site until it is resolved.

Trim the strings of the IUD to 3-4 cm in length and note the string length. Avoid cutting the strings too short. If the client or her partner becomes aware of the threads, they may be cut shorter in length at the follow-up visit.

Remove the speculum and assess the woman.

DETAILED DESCRIPTION:
Only clinicians with proven proficiency in IUD insertion will be allowed to perform insertions . The steps of the IUD insertion procedure will be explained to the woman.

Perform a bimanual examination to determine the size, shape, and position of the uterus.

Insert a warm, moistened speculum. Cleanse the cervix with an antiseptic solution using 3 scoppettes or more (one for each sweep of the cervix).

Open the sterile insertion instruments without touching the inside of the packet and place within easy reach.

Remove the tenaculum by its handle and grasp the anterior or posterior lip of the cervix. Close gently to the first notch. Having the woman to cough while the tenaculum is being attached can ease the pinch.

Apply gentle traction with the tenaculum to straighten the canal. Remove the sound by its handle and gently insert to measure the depth of the uterus. Do not apply great force if there is resistance. Apply further traction to the tenaculum and attempt to re-insert the sound at a different angle. Once the sound is inserted and removed, note the depth of the uterine cavity. The woman can expect to feel cramping as the sound is inserted and withdrawn.

Open the IUD pack without touching its contents. Put on sterile gloves. Load the IUD and insert it into the uterine cavity according to the manufacturer instructions. As the IUD is inserted through the cervix into the uterus, the patient may have pain and cramping similar to strong menstrual cramps.

Gently remove the tenaculum. Tamponade any bleeding from the tenaculum site until it is resolved.

Trim the strings of the IUD to 3-4 cm in length and note the string length. Avoid cutting the strings too short. If the client or her partner becomes aware of the threads, they may be cut shorter in length at the follow-up visit.

Remove the speculum and assess the woman.

ELIGIBILITY:
Inclusion Criteria:

* 1. Multiparous women from 20 - 40 years of age , seeking contraception and choosing IUD as their preferred method after proper and thorough counseling.

  2. Regularly menstruating women ( menstural cycle varying between 24- 38 days).

  3. Contraceptive pills or any type of hormonal medication had not been taken for at least 3 months prior to the study, and any IUD had necessarily been removed at least 3 months earlier.

Exclusion Criteria:

* • Pregnancy or suspicion of pregnancy

  * Congenital or acquired uterine anomalies which distort the uterine cavity (fibroids, endometrial polyps, cervical stenosis, bicornuate uterus, small uterus < 6 cm)
  * Acute PID or a history of PID within the past 3 months
  * Postpartum or post-abortion endometritis within the past 3 months
  * Current STI or within the past 3 months (including cervicitis)
  * Cervical cancer
  * Endometrial cancer
  * Malignant gestational trophoblastic disease
  * Undiagnosed vaginal bleeding
  * Hypersensitivity to any component in the IUD (copper, progesterone)
  * Less than 4 weeks postpartum.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 300 (Actual)
Dates: Start 2019-12-02 (Actual); Primary Completion 2021-08-11 (Actual); Study Completion 2021-08-11 (Actual)

PRIMARY OUTCOMES:
menorrhagia | 6 months after IUD insertion
  occurrence of heavy menstrual flow

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed maged, Study Director — professor
Locations (1):
- Kasr Alainy medical school, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No